CLINICAL TRIAL: NCT07188324
Title: Fetal Kidney Length and Gestational Age in Late 2nd and 3rd Trimesters
Brief Title: Assessment of Mean Fetal Kidney Length as a Reliable Parameter for Accurate Estimation of Gestational Age in Late 2nd and 3rd Trimesters
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mostafa Mohammed Refaay El shemy, Assistant professor of Obstetrics and Gynecology faculty of medicine, Cairo University
Other Study IDs: Fetal kidney length by 2D us
Record Dates: First submitted 2025-09-12; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fetal Conditions
Keywords: Fetal kidney - length-gestational age -2D- ultrasound

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Accurate GA estimation is necessary when early termination of pregnancy is necessary as soon as the fetus becomes mature e.g. cases of pre-eclampsia, chronic renal disease, severe intrauterine growth retardation (IUGR), diabetes and placenta praevia centralis. Accurate GA estimation is also necessary where certain tests need to be performed for example amniotic fluid and serum assays, chorionic villus sampling and to plan fetal therapies. (Gupta DP et al., 2013)

DETAILED DESCRIPTION:
There are number of parameters used to calculate gestational age, but the most commonly used by all sonologists is a composite gestational age obtained by biparietal diameter (BPD), head circumference (HC), abdominal circumference (AC), and femur length (FL) in the second and third trimesters (Jae SS et al., 2007). Even these may not provide gestational age with great accuracy owing to discrepancies in late-trimester scans and intrauterine growth restriction (IUGR).

Fetal kidney shows steady growth of 1.1 mm/ gestational week throughout the pregnancy unaffected by any underlying growth abnormalities (Ahmadi et al., 2015). By prenatal ultrasound, identification of either one or both kidneys is possible in 90% of cases in the 17th week of gestation and in 95% of cases after the 20th week. Although kidney size, as for all fetal organs, is affected by growth variations, these appear to predominantly affect only anterior- posterior and transverse diameters (width of kidney) (Callen A., 2008). However, its length shows no significant change with any underlying medical condition (Kansaria and Parulekar, 2010).Fetal kidney length (FKL) has recently been found to have a strong correlation with gestational age. According to the investigations, the fetal kidney length may be utilized to estimate gestational age when dates are ambiguous or when women seek ultrasound fetal biometry dating during the third trimester itself (Kansaria J et al., 2009). Fetal kidney length (FKL), according to a number of studies, closely corresponds with gestational age in the third trimester. Although ultrasound textbooks frequently include tables of various sizes, the fetal kidney has not received much research as a biometric criterion for estimating gestational age(Goyal L et al., 2016).

This study aims to assess the uses of the mean fetal kidney length as reliable parameter for accurate determination of gestational age in late 2nd and/or 3rd trimesters (24 weeks - 40 weeks) in cases who are not sure about their last menstrual period and need proper management of any health problem such as preeclampsia, diabetes or fetal growth abnormality.

ELIGIBILITY:
Inclusion Criteria:

* All healthy women with viable normal singleton pregnancies in their late second and third trimesters (24 weeks - 40 weeks) calculated from their last menstrual period.
* Women who will sure of the dates of their last menstrual period (1st day) and/or those with first obstetrics dating using crown rump length (CRL). 3- Women with regular menstrual cycle in last three months before their last menstrual period.

Exclusion Criteria:

* Women with high-risk pregnancies such as preeclampsia, diabetes, hypertension, polyhydramnios.

  ❖ Maternal:
* Multiple pregnancies.
* Gross maternal obesity.

  ❖ Fetal:
* Fetus with congenital anomalies especially renal anomalies.
* Fetuses with abnormal renal morphology (a genesis, hypoplasia, cysts, nephromegaly, polycystic kidney, hydronephrosis, etc.…
* Fetuses with renal pelvic dilatation of 5 mm or greater, obscured adrenal and renal border.
* Fetus with growth abnormalities (intrauterine growth retardation or macrosomia).

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Healthy pregnant women at their late second and third trimester by reliable LMP who will meet the inclusion criteria, attend the fetal medicine Unit at Cairo University Hospital and consent to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of estimation of mean fetal kidney length in comparison with other parameters | 18months
  Estimation of the gestational age (GA) in weeks by measurement of mean fetal kidney length (MFKL)in mm and detect its accuracy in correlation with gestational age derived from other traditional fetal parameters (BPD, HC, AC& FL) in mm and actual gestational age derived from first day of last menstrual period.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo University, Giza, Cairo Governorate, Egypt